CLINICAL TRIAL: NCT00390390
Title: A Phase III, Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group Trial of 14 Day Treatment With Lansoprazole 15 mg Once a Day in Frequent Heartburn
Brief Title: Efficacy/Safety of Lansoprazole in Patients With Frequent Heartburn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRSW-GN-302
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2007-04

CONDITIONS: Heartburn
Keywords: Heartburn, frequent heartburn, proton pump inhibitor, lansoprazole
MeSH Terms: conditions — Heartburn | interventions — Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole

SUMMARY:
Heartburn, a burning sensation in the chest or throat, occurs in many patients when acidic stomach contents move into the esophagus from the stomach. This study will investigate the safety and efficacy of lansoprazole 15 mg once a day in treating frequent heartburn.

ELIGIBILITY:
Inclusion Criteria:

1. Experiencing heartburn at least 2 days per week over the past month.
2. Having heartburn that responds to heartburn medication.
3. Be willing to discontinue the use of heartburn treatment for 7 days prior to inclusion in the study.

Exclusion Criteria:

1. Having history of erosive esophagitis or gastroesophageal reflux disease diagnosed by a physician and confirmed by testing (endoscopy).
2. Be unwilling to take only the study medication, and antacid provided as a rescue medication for relief of acute heartburn during the study.

Other protocol-defined inclusion or exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576
Dates: Start 2006-06; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate that repeated daily doses of 15 mg of lansoprazole are effective in increasing the proportion of days with no heartburn during study treatment, when compared to placebo.

SECONDARY OUTCOMES:
To determine the proportion of nighttimes with no heartburn during 14 days of treatment in subjects receiving lansoprazole versus placebo
To determine the proportion of subjects with no heartburn during day 1 in those receiving lansoprazole versus placebo
Evaluation of lansoprazole safety.

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Sunbelt Research Group, Mobile, Alabama
  - Arkansas Primary Care Clinic, Little Rock, Alaska
  - Radiant Research, Chandler, Arizona
  - Radiant Research - Scottsdale, Scottsdale, Arizona
  - Edinger Medical Group, Fountain Valley, California
  - Gaslamp Medical Center, San Diego, California
  - Expresscare Clinical Research, Colorado Springs, Colorado
  - Central Florida Clinical Trials inc., Altamonte Springs, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Health Awareness Inc., Jupiter, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Palm Beach Research, West Palm Beach, Florida
  - Accelovance, Peoria, Illinois
  - IRSI, Rockland, Massachusetts
  - Prime Care Research, St Louis, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Urgentmed, South Bound Brook, New Jersey
  - Wake research associates, Inc, Raleigh, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Radiant Research, Cincinnati, Ohio
  - Wells Institute For Health Awareness, Kettering, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Durham Physicans, Durham, Pennsylvania
  - 2222 State Street, Nashville, Tennessee
  - Wells Branch Medical Center, Austin, Texas
  - Medical Edge Healthcare Group, Dallas, Texas
  - Houston, Texas
  - Clinical Trials Network, Houston, Texas
  - Health Research of Hampton Roads, Newport News, Virginia
  - Holston Medical Group, Weber City, Virginia